CLINICAL TRIAL: NCT05536297
Title: An Open-label Extension (OLE) Phase 3 Trial to Assess the Safety of Intravitreal Administration of Avacincaptad Pegol (Complement C5 Inhibitor) in Patients With Geographic Atrophy Who Previously Completed Phase 3 Study ISEE2008 (GATHER2)
Brief Title: Avacincaptad Pegol Open-Label Extension for Patients With Geographic Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISEE2009; 2022-002860-59 (EudraCT Number); 2024-515185-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: Geographic Atrophy;; Macular Degeneration;; ARC1905;; Avacincaptad pegol;; Zimura (previous name);; Izervay
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- avacincaptad pegol (Experimental): Participants will receive avacincaptad pegol 2 mg monthly from Month 1 to Month 17.
  Interventions: Drug: avacincaptad pegol

INTERVENTIONS:
Drug: avacincaptad pegol — Intravitreal Injection
  Other Names: Zimura (previous name); ARC1905; Izervay

SUMMARY:
The purpose of this study is to assess long-term safety of avacincaptad pegol intravitreal administration for patients with geographic atrophy (GA) who completed Study ISEE2008 (GATHER2) through the Month 24 visit on study treatment (either avacincaptad pegol or Sham).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 50 years or greater diagnosed with GA inside and/or outside of the fovea who completed Study ISEE2008 (GATHER2) through the Month 24 visit on study treatment.
* Patient must provide new written informed consent for this OLE trial prior to participation.
* Patient must have the ability to return for all trial visits for the duration of the 18-month trial.

Exclusion Criteria:

* Patient did not complete Study ISEE2008 (GATHER2) through the Month 24 visit on study treatment (either avacincaptad pegol or Sham),
* Patient who had the study drug permanently withdrawn for an AE during ISEE2008 are not eligible.
* Patient did not enroll into this OLE trial within the 90 day enrollment period.
* Patient who is pregnant or nursing

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 18 Months
  An AE is defined as any untoward medical occurrence in a participant including unfavorable and unintended signs, symptoms or disease temporally associated with the use of a medicinal product and which does not necessarily have to have a causal relationship to this treatment.
  AEs include illnesses with onset during the trial, or exacerbations of pre-existing illnesses. Exacerbation of pre existing illness is defined as a significant increase in the severity of the illness as compared to the start of the trial and should be considered when a participant requires new or additional treatment for that illness.

SECONDARY OUTCOMES:
Number of participants with Anti-Drug Antibody (ADA) status | Up to 18 Months
  ADA will be recorded from the serum samples collected. Overall ADA status will be reported: ADA-negative, ADA positive, ADA-inconclusive and unevaluable sample.
Pharmacokinetics (PK) of avacincaptad pegol in plasma: concentration | Up to 18 Months
  Concentration will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (117):
- United States (53):
  - Retinal Diagnostic Center, Campbell, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - Jacobs Retina Center at The Shiley Eye Institute USCD, La Jolla, California
  - Jules Stein Eye Institute David Geffen School of Medicine, Los Angeles, California
  - Doheny Eye Center, UCLA, Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Orange County Retinal Med Group, Santa Ana, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern CO, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Center for Retina & Macula Disease, Winter Haven, Florida
  - Southeast Retina Center P.C., Augusta, Georgia
  - Retina Consultants of Hawaii, Inc., ‘Aiea, Hawaii
  - Illinois Eye Center, Peoria, Illinois
  - Vitreo Retinal Consultants & Surgeons, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Research Institute at New England Retina, Springfield, Massachusetts
  - Vitreoretinal Associates PC, Worcester, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Retina Vitreous Surgeons of Central New York, Liverpool, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Retina Associates of Western NY, Rochester, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Retina & Vitreous Center of Southern Oregon, PC, Ashland, Oregon
  - Retina Northwest PC, Portland, Oregon
  - Eye Health Northwest, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Institute, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Retina Research of Beaufort, Beaufort, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Retina Research Institute of Texas, LLC, Abilene, Texas
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah PC, Salt Lake City, Utah
  - Pacific Northwest Retina, Bellevue, Washington
- Argentina (5):
  - Oftalmólogos Especialistas, Rosario, Sante Fe
  - Centro Oftalmológico Dr. Charles, Buenos Aires
  - Instituto Oftalmologico de Buenos Aires, Buenos Aires
  - Oftar Mendoza, Mendoza
  - Microcirugia Ocular, Santa Fe
- Australia (2):
  - Centre for Eye Research Australia, East Melbourne
  - Sydney Retina Clinic, Sydney
- Austria (3):
  - Medizinische Universitat Graz, Styria
  - Medizinische Universitat Innsbruck, Tyrol
  - Medical University of Vienna, Department of Ophthalmology and Optometry, Vienna
- Centre H. U. Brugmann, Brussels, Belgium
- Brazil (3):
  - Centro de Ensino e Pesquisa do Instituto de Visao, Belo Horizonte
  - Universidade Federal de Sao Paulo, São Paulo
  - IPEPO - Instituto da Visao, São Paulo
- Canada (3):
  - Calgary Retina Consultants, Calgary, Alberta
  - St. Joseph's Health Care London, London, Ontario
  - Retina Centre of Ottawa, Ottawa, Ontario
- Colombia (2):
  - Fundacion Oftalmologica Nacional, Bogotá
  - Clinica de Oftalmologia Sandiego, Medellín
- Clinical Hospital Osiiek, Ophthalmology Clinic, Osijek, Croatia
- Lékárna nad Knížecí Kováků, Smíchov, Czechia
- France (11):
  - University Hospital of Bordeaux, Bordeaux
  - Hopital Intercommunal de Creteil, Créteil
  - Pole Vision Val D'Ouest, Écully
  - Centre Ophtalmologique Rabelais, Lyon
  - Hopital de la Croix-Rousse, Lyon
  - Centre Paradis-Monticelli, Marseille
  - Centre D'exploration Ophtalmologique De L'odéon, Paris
  - Centre d'Imagerie et Laser, Paris
  - Rothschild Foundation, Paris
  - Hopital Lariboisiere, Service Pharmacie, Paris
  - Centre Ophtalmologique Saint Exupéry, Saint-Cyr-sur-Loire
- Germany (5):
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinik für Augenheilkunde, Medizinische Hochschule Hannover, Hanover
  - Augenklinik der Ludwig-Maximilian Universität München, München
  - Eye Clinic Ludwig Maximilian, München
  - Augenzentrum am St. Franziskus-Hospital, Münster
- Hungary (3):
  - Dept. of Ophthalmology Semmelweis University Budapest, Budapest
  - Bajcsy Zsilinszky Korhaz Szemeszet, Budapest
  - Budapest Retina Associates, Budapest
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
  - Kaplan Medical Center, Rehovot
  - Shamir Medical Center, Tzrifin
- Italy (9):
  - AOU Policlinico S. Orsola-Malpighi, Bologna
  - Clinica Oftalmologica Ospedale C. S.S. Annunziata, Chieti
  - Ospedaliero Universitaria di Ferrara, Ferrara
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Fatebenefratelli, Milan
  - Azienda Ospedaliera U. della Campania "Vanvitelli", Napoli
  - Policlinico Tor Vergata, Roma
  - Azienda Ospedaliero-U.Ospedali Riuniti Umberto I, Torrette Di Ancona
- P. Stradins Clinical university hospital, Riga, Latvia
- Spain (10):
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Clinicade Oftalmologia Barraquer, Barcelona
  - Institut Catala de la Retina, Barcelona
  - Instituto Clinico Quirurgico de Oftalmologia, Bilbao
  - Hospital La Arruzafa, Córdoba
  - Valles Ophthalmology Research (VOR) in Hospital General de Catalunya Pedro, Sant Cugat del Vallès
  - Instituto Oftalmológico Gómez-Ulla, Santiago de Compostela
  - IMED Servicio Oftalmología, Valencia
  - Rio Hortega University Hospital, Valladolid
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/